CLINICAL TRIAL: NCT02725840
Title: Early Markers of Subclinical Pulmonary Vascular Radiation Toxicity in Breast Cancer
Brief Title: Breast Cancer Lung Late Effects
Acronym: BELLE
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Collaborators: Florida Department of Health (Other Government)
Responsible Party: Sponsor
Other Study IDs: IRB201600387; OCR14962 (Other: UF OnCore); 6BC09 (Other Grant/Funding Number: FL DEPT OF HLTH BANKHEAD-COLEY CANCER RE)
Record Dates: First submitted 2016-03-21; First posted 2016-04-01 (Estimated); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Radiation Injury; Breast Cancer
Keywords: pulmonary vasculature; radiation late effects; proton therapy
MeSH Terms: conditions — Radiation Injuries; Breast Neoplasms | interventions — Proton Therapy; Respiratory Physiological Phenomena

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood plasma collection
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Proton beam radiation therapy: The participants in this group will be receiving proton therapy of the affected breast and chest wall as part of their standard of care. In addition, a Computed Tomography (CT) Scan of the chest wall will be performed, and pulmonary function test (PFT).
  Interventions: Radiation: Proton beam radiation therapy.; Procedure: Computed Tomography (CT) Scan; Procedure: Pulmonary Function Test (PFT)
- X-ray based radiation therapy: The participants in this group will be receiving X-ray radiation therapy of the affected breast and chest wall as part of their standard of care. In addition, a Computed Tomography (CT) Scan of the chest wall will be performed, and pulmonary function test (PFT).
  Interventions: Radiation: X-ray based radiation therapy; Procedure: Computed Tomography (CT) Scan; Procedure: Pulmonary Function Test (PFT)

INTERVENTIONS:
Radiation: Proton beam radiation therapy. — Proton bean radiation therapy interact differently with tissue with the result that protons are absorbed completely within the tissue instead of primarily passing through the entire body. The maximal depth of penetration is dependent upon the incoming velocity (energy) of the protons. Proton therapy utilizes this property to deliver radiation with very little dose beyond the targeted lesion. The dose-rate will be managed as part of the standard of care.
  Other Names: PTI
  Groups: Proton beam radiation therapy
Radiation: X-ray based radiation therapy — The three-dimensional (3D) mapping of radiation dose distributions permits detailed assessment of local vascular damage as a function of treatment factors of dose, dose-rate. The dose-rate will be managed as part of the standard of care.
  Other Names: conformal RT
  Groups: X-ray based radiation therapy
Procedure: Computed Tomography (CT) Scan — Computed Tomography (CT) Scan of the chest will be performed at 1, 3, 6, 12, 18 and 24 months
Procedure: Pulmonary Function Test (PFT) — Pulmonary function test (PFT) will be performed at pre-treatment, and at 6 and 12 months.

SUMMARY:
Through improved early detection and treatment, the number of long term breast cancer survivors continues to increase. There are now 2.8 million breast cancer survivors in the U.S. Florida alone adds over 9,000 women to the survivorship pool each year. Most receive radiation treatment (RT) of the affected breast and chest wall to reduce risk of recurrence. Even with advanced radiation techniques for dose conformality to minimize exposure of the highly sensitive lung, 14% of breast cancer patients treated with radiation develop clinical pulmonary toxicity, with 4% overall experiencing high grade clinical toxicity. Early diagnosis and intervention to mitigate lung radiation toxicity is increasingly important for the long term care of these survivors.

The investigators' goal is to better identify breast cancer patients at high risk for experiencing severe pulmonary toxicity requiring medical intervention, provide a means to identify toxicity early on, and tailor treatment and/or early intervention on a per-patient basis.

DETAILED DESCRIPTION:
This project involves repeat chest computed tomography (CT) imaging and blood draws in subjects with breast cancer with radiation treatment to the affected breast and chest wall. The investigators are studying women receiving one of 2 types of radiation, either conventional X-rays (IMRT) or protons at the University of Florida Health Proton Therapy Institute (UFHPTI). These subjects typically would not receive follow-up chest CTs as per standard of care. All subjects will have received a pre-treatment chest CT scan as part of the treatment planning process. The investigators will enroll 30 subjects in the X-ray treatment group and 25 subjects in the proton group.

The investigative team has recently solved the technical challenges of extracting and characterizing lung vascular anatomy from clinical CT images of the chest and used these tools to characterize acute and chronic changes to pulmonary vascular structure in breast cancer patients receiving radiation to the chest wall for treatment of their cancer.

In Aim 1 of this study the investigators will compare lung vascular damage in women treated with conventional radiation with those treated at the UFHPTI. In Aim 2 they will use blood samples of the subjects of Aim 1 to investigate the differential role of inflammatory cytokines in the initiation and progression of pulmonary vascular radiation response in conventional versus proton radiation exposures. Aim 3 compares vascular damage with clinical pulmonary function assessment using spirometry and diffusion capacity of carbon monoxide (DLCO). Aim 4 ties together Aims 1-3 by employing and extending existing mathematical models of radiobiological response to improve and solidify the scientific understanding of the biological mechanisms of radiation response.

ELIGIBILITY:
Inclusion Criteria:

* Women who are at least 18 years of age.
* Women with Stage II or higher primary breast cancer and who are scheduled to receive conventional X-ray RT (n=30) or proton therapy (n=25) to the breast and chest wall.

Exclusion Criteria:

* Patients not willing or able to submit to repeat chest CT scans and blood draws.
* Pregnant women.
* Patients who have previously had radiation treatment where any portion of the lung received greater than 5 Gy of radiation exposure.
* Women with bilateral breast cancer or metastatic disease to sites near the chest where additional radiation exposure to any portion of the lung of greater than 5 Gy is anticipated.
* Women with allergic reaction to all common CT contrast agents.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients who are 18 years of age or older and have Stage II or higher disease and who are scheduled to receive conventional X-ray RT (n=30) or proton therapy (n=25) to the breast and chest wall for the treatment of breast cancer will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2022-01-14 (Actual); Study Completion 2022-01-14 (Actual)

PRIMARY OUTCOMES:
The lower dose limit for measurable change in number of small blood vessels as characterized from chest CT scans at 1,3,6, 12 and 24 months (= 2 years) and compared between proton versus X-ray radiation therapy. | 2 years
  The investigators seek to identify differences between the treatment modalities (proton versus X-ray) in regards to the lower dose limits for change in number of small blood vessels as measured from chest CT scans and quantified using the team's analysis technique.
Vessel number change dose-response relationship as measured from chest CT scans at 1,3,6, 12 and 24 months (= 2 years) and compared between proton versus X-ray radiation therapy. | 2 years
  Identify change in number of small blood vessels as measured from chest CT scans and quantified using the team's analysis technique, as a function of radiation dose exposure across the lung.
Recovery of number of small blood vessels as measured from chest CT scans acquired at 1,3,6, 12 and 24 months (= 2 years) and compared between proton versus X-ray radiation therapy. | 2 years
  Identify differences in temporal patterns of vessel regeneration following radiation exposure as a function of dose and of modality (proton versus X-ray).
Temporal patterns of blood cytokines following radiation exposure as measured from blood draws a pre-treatment and at 1,3,6, 12 and 24 months (= 2 years), and compared between proton versus X-ray radiation therapy. | 2 years
  Quantify differences in temporal patterns of levels of cytokines in the blood in breast cancer patients receiving conventional X-ray versus proton RT using serial blood draws that are time-matched with the CT chest scans.
Correlate change in number of small blood vessels as measured from chest CT scans at 1,3,6, 12 and 24 months (= 2 years) with clinical pulmonary function test outcomes at 6 and 12 months. | 1 year
  Correlate change in number of small blood vessels as measured from chest CT scans and quantified using the team's analysis technique, with clinical pulmonary function test (spirometry and diffusion capacity for carbon monoxide) outcomes to identify potential predictive value of early vascular changes to conventional clinical measures of late effects.

SECONDARY OUTCOMES:
Compare incidence of long-term clinical grade 2 and higher radiation toxicity to the lung as documented in patient medical records and compared between proton versus X-ray radiation therapy. | 8 years
  The goal is to monitor long-term (>8 year) incidence of clinical pulmonary toxicity in these subjects to identify any difference between X-ray and proton treatment methodologies.
Compare duration of overall survival and whether death was attributed to lung radiation toxicity as documented in patient medical records and compared between proton versus X-ray radiation therapy. | 8 years
  The goal is to monitor long-term (>8 year) survival in these subjects to identify any difference between X-ray and proton treatment methodologies.

OTHER OUTCOMES:
Document patterns of metastatic presentation as observed from chest CT scans at 1,3,6, 12 and 24 months (= 2 years). | 2 years
  To identify patterns of asymptomatic metastatic progression in those subjects who develop recurrence to the thorax during the follow-up imaging period,

CONTACTS AND LOCATIONS:
Overall Officials: Walter O'Dell, PhD, Principal Investigator — University of Florida; Julie Bradley, PhD, Principal Investigator — University of Florida
Locations (2):
- United States (2):
  - Department of Radiation Oncology Davis Cancer Pavilion, Gainesville, Florida
  - University of Florida Health Proton Therapy Institute, Jacksonville, Florida

IPD SHARING:
Plan to Share IPD: Undecided